CLINICAL TRIAL: NCT07009964
Title: AI-Enhanced Educational Intervention to Support Contextual Well-being in Young Adults (ContextWell)
Brief Title: An Exploratory Feasibility Study
Acronym: Contextwell
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: UCD Clinical Research Centre, Ireland (Unknown); University College Cork (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ContextWell-2025
Record Dates: First submitted 2025-05-07; First posted 2025-06-08 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Well-Being; Lifestyle, Healthy; Young Adult; Behavior and Behavior Mechanisms
Keywords: Student well-being; Artificial Intelligence; Contextual Well-being; Contextual AI; Preventive health; Digital Health; Lifestyle medicine; Pilot study; Proof of concept
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ContextWell Educational Programme (Other): Participants will engage in the ContextWell programme, an online well-being education intervention that supports the development of core meta-skills such as self-awareness, reflective thinking, and value-based decision-making. These skills help participants take ownership of their well-being and support their ability to independently pursue and apply knowledge that promotes health. This includes, for example, adopting principles related to lifestyle medicine such as stress management, sleep improvement, nutrition, and physical activity. The programme does not teach lifestyle medicine directly. Instead, it builds the foundational mindset and capacities that enable participants to seek out and integrate such practices into their lives and future clinical roles.
  Interventions: Other: ContextWell Educational Programme

INTERVENTIONS:
Other: ContextWell Educational Programme — ContextWell Educational Programme

SUMMARY:
This study explores the feasibility of ContextWell, a well-being education programme that combines an online webinar with an AI-powered behavioural nudging system. The programme aims to support university students, particularly those in healthcare disciplines, in enhancing well-being and adopting healthier lifestyle habits.

The primary objective is to determine whether the programme can be feasibly delivered within university settings. A secondary objective is to assess its potential to improve student well-being and encourage behavioural changes aligned with lifestyle medicine principles.

The intervention builds on the understanding that healthcare professionals' lifestyle habits and well-being have a direct impact on patient care. Focusing on healthcare students helps advance the integration of lifestyle medicine within health education and clinical practice.

This single-group feasibility study delivers the full intervention to all participants. Students participate in an online well-being webinar and receive AI-generated behavioural prompts designed to promote self-awareness and healthier daily choices.

Key evaluation measures will indicated the feasibility of the programme among young adults in academic environments. Participant feedback and initial outcomes will support future development and inform larger-scale research.

ELIGIBILITY:
Inclusion Criteria:

Primarily healthcare students, young adults enrolled in higher education (18-30 years old)

Access to a computer or mobile device with an internet connection;

Willingness to participate in the educational webinar;

Willingness to complete AI-driven assignments;

Able to read and understand English.

Exclusion Criteria:

Are under the age of 18, or above 30;

Inability to access a computer or mobile device with internet connection;

Inability to read or understand English;

Unwillingness to participate in the webinar or complete assignments.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Up to 4 weeks post-study launch (enrolment period).
  Description: Proportion of eligible participants who enroll in the ContextWell Programme.
  Metric: % of enrolled participants out of those approached.
  Measurement Method: Screening and enrolment logs.
Retention Rate | Through study completion, an average of 5 weeks post-baseline.
  Proportion of enrolled participants completing the programme.
  Metric:
  1. % completing final follow-up.
  2. Count completing all study components.
  Measurement Method: Attendance records, programme tracking data, follow-up survey.

SECONDARY OUTCOMES:
Acceptability of the Intervention | At 2 weeks post-intervention.
  Description: Participants' satisfaction with the content, format, and delivery.
  Metric: Mean satisfaction rating; qualitative feedback.
  Measurement Method: Post-intervention survey (Likert-scale + open-ended items).
Demand for the Programme | At 2 weeks post-intervention.
  Participants' expressed interest in continued use and peer recommendation.
  Metric: % intending to continue use or recommend.
  Measurement Method: Survey responses on future use/recommendation.
Implementation Feasibility | During intervention period, Weeks 1 to 3 post-baseline.
  Practicality of delivering the intervention as planned.
  Metric: Number of technical issues.
  % of content delivered as intended.
  Measurement Method: Researcher logs, participant feedback.
Perceived Impact on Well-Being | At 4 weeks post-baseline.
  Participants' perception of effects on well-being
  Metric: % reporting improved well-being.
  Measurement Method: follow-up survey (Likert-scale and reflections).

CONTACTS AND LOCATIONS:
Overall Officials: Walter Prof. Cullen, MD, Study Chair — University College Dublin
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No